CLINICAL TRIAL: NCT04587687
Title: A Phase II Study of Brentuximab Vedotin Plus Bendamustine for Relapsed/Refractory Follicular Lymphoma
Brief Title: Brentuximab Vedotin and Bendamustine for the Treatment of Relapsed or Refractory Follicular Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Joseph Tuscano (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Seagen Inc. (Industry)
Responsible Party: Sponsor-Investigator, Joseph Tuscano, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC#284; NCI-2020-06645 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCDCC#284 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH)
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Recurrent Follicular Lymphoma; Refractory Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Bendamustine Hydrochloride; Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (brentuximab vedotin, bendamustine) (Experimental): Patients receive brentuximab vedotin IV over 30 minutes on day 1 and bendamustine IV over 60 minutes on days 1 and 2. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients who respond to combination treatment and do not experience excessive toxicity may continue to receive brentuximab vedotin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 10 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bendamustine Hydrochloride; Drug: Brentuximab Vedotin

INTERVENTIONS:
Drug: Bendamustine Hydrochloride — Given IV
  Other Names: Bendamustin Hydrochloride; Bendeka; Cytostasan Hydrochloride; Levact; Ribomustin; SyB L-0501; Treanda
Drug: Brentuximab Vedotin — Given IV
  Other Names: ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; cAC10-vcMMAE; SGN-35

SUMMARY:
This phase II trial investigates how well brentuximab vedotin and bendamustine work in treating patients with follicular lymphoma that has come back (relapsed) or does not respond to treatment (refractory). Brentuximab vedotin is a monoclonal antibody, brentuximab, linked to a toxic agent called vedotin. Brentuximab attaches to CD30 positive cancer cells in a targeted way and delivers vedotin to kill them. Chemotherapy drugs, such as bendamustine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. This trial is being done to determine if the combination of brentuximab vedotin plus bendamustine is safe and to determine the effectiveness of the combination.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Obtain a preliminary estimate of the anti-tumor activity of brentuximab vedotin plus bendamustine hydrochloride (bendamustine) in patients with relapsed/refractory (R/R) CD30+ follicular lymphoma as determined by the complete response rate (CR) and best overall response rate (ORR) as defined per Lugano criteria.

SECONDARY OBJECTIVES:

To obtain the duration of response (DOR). To obtain the time to response (TTR). To obtain the progression-free survival (PFS) among subjects with relapsed or refractory CD30-positive follicular lymphoma (FL) receiving brentuximab vedotin and bendamustine. To obtain data on overall survival (OS). To evaluate the safety and tolerability.

OUTLINE:

Patients receive brentuximab vedotin intravenously (IV) over 30 minutes on day 1 and bendamustine IV over 60 minutes on days 1 and 2 of each cycle. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients who respond to combination treatment and do not experience excessive toxicity may continue to receive additional single-agent brentuximab vedotin IV over 30 minutes on day 1 (once every 21 days) for up to 10 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days, and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed relapsed or refractory follicular CD30+ non-Hodgkin lymphoma (NHL) (included in this category are follicular grade I, II, IIIa). CD30 positivity > 1% (tumor cells or surrounding peripheral microenvironment)
* Patients must have measurable disease by computed tomography (CT) or positron emission tomography (PET) scan, with one or more sites of disease >= 1.5 cm in longest dimension
* Relapsed or refractory disease after at least 1 prior regimen, defined using the 2014 Lugano classification
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 3 months
* Leukocytes >= 2,500/mcL
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 50,000/mcL
* Hemoglobin >= 8 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (however, patients with known Gilbert disease who have serum bilirubin level =< 3 x ULN may be enrolled)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN (AST and/or ALT =< 5 x ULN for patients with liver involvement)
* Alkaline phosphatase =< 2.5 x ULN (=< 5 x ULN for patients with documented liver involvement or bone metastases)
* Creatinine clearance >= 30 mL/min/1.73 m^2 by Cockcroft-Gault
* Institutional normalized ratio (INR) and partial thromboplastin time (aPTT) =< 1.5 x ULN (This applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation, such as low-molecular-weight heparin or warfarin, should be on a stable dose.)
* Administration of bendamustine or brentuximab vedotin may have an adverse effect on pregnancy and poses a risk to the human fetus, including embryo-lethality. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 5 months (150 days) after the last dose of study agent. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Patients positive for human immunodeficiency virus (HIV) are allowed on study, but HIV-positive patients must have:

  * A stable regimen of highly active anti-retroviral therapy (HAART)
  * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
  * A CD4 count above 250 cells/mcL and an undetectable HIV viral load on standard polymerase chain reaction (PCR)-based tests

Exclusion Criteria:

* Patients who have had chemotherapy, or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C, steroid treatment for follicular lymphoma is allowed per protocol) prior to entering the study or those who have not recovered from adverse events (other than alopecia) due to agents administered more than 2 weeks earlier. Specifically, the following therapies are not allowed:

  * Herbal therapy (1 week washout required)
  * Treatment with any other investigational agent within 3 weeks prior to cycle 1, day 1.
  * Prior therapy with bendamustine or a bendamustine-containing regimens with progression within 6 months of receiving treatment
* Current or prior use of immunosuppressive medications (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 14 days prior to first dose (cycle 1, day 1). The following are exceptions to this criterion:

  * Intranasal, inhaled, topical or local steroid injections (e.g., intra-articular injection); steroids as premedication for hypersensitivity reactions; systemic corticosteroid at physiologic doses not to exceed 10 mg/day of prednisone or equivalent may be enrolled
  * Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled
  * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
  * Patients taking bisphosphonate therapy for symptomatic hypercalcemia. Use of bisphosphonate therapy for other reasons (e.g., bone metastasis or osteoporosis) is allowed
* Patients with known uncontrolled central nervous system (CNS) involvement by lymphoma, including leptomeningeal involvement
* History of hypersensitivity to bendamustine or brentuximab vedotin or any excipient
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to other agents used in study
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease.

  * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible.
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA)
* Neuropathy grade > 1
* Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

  * Rash must cover less than 10% of body surface area (BSA)
  * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%)
  * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* Patients with known active tuberculosis (TB) are excluded
* Severe infections within 4 weeks prior to cycle 1, day 1, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection within 2 weeks prior to cycle 1, day 1
* Received oral or intravenous (IV) antibiotics within 2 weeks prior to cycle 1, day 1. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible
* Major surgical procedure within 28 days prior to cycle 1, day 1 or anticipation of need for a major surgical procedure during the course of the study
* Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine within 4 weeks prior to cycle 1, day 1 or at any time during the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2020-12-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate | Up to 2 years
  Will be assessed per 2014 Lugano criteria and Lymphoma Response to Immunomodulatory Therapy Criteria (LYRIC) criteria. Will be summarized with 95% confidence intervals.
Best overall response rate (ORR) | Up to 2 years
  Will be assessed by complete response + partial response per 2014 Lugano criteria and LYRIC criteria.

SECONDARY OUTCOMES:
Duration of response | From time of initial response assessment demonstrating at least partial response until disease response assessment that demonstrates progressive disease, assessed up to 2 years
  Will be summarized descriptively using the Kaplan-Meier estimate.
Time to response | From registration to first disease response assessment that demonstrates at least partial response, assessed up to 2 years
  Will be summarized descriptively using the Kaplan-Meier estimate.
Progression-free survival | From registration until death, relapse/progression, receipt of anti-lymphoma therapy, or last follow-up, whichever comes first, assessed up to 2 years
  Disease relapse/progression will be defined according to the 2014 International Harmonization Project (IHP) criteria. Will be summarized descriptively using the Kaplan-Meier estimate.
Overall survival | From registration to death due to any cause, assessed up to 2 years
  Will be summarized descriptively using the Kaplan-Meier estimate.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Tuscano, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States